CLINICAL TRIAL: NCT00495482
Title: Incurable Ill Patients Attitudes to Euthanasia and Assisted Suicide: A Prospective, Multi-Centre Trial in Palliative Care Units in Saxony
Brief Title: Incurable Ill Patients Attitudes Towards Euthanasia and Assisted Suicide
Acronym: ESPIL
Status: Completed | Type: Observational
Sponsor: Klinikum St. Georg gGmbH (Other)
Responsible Party: Principal Investigator, Armin Sablotzki, MD, Prof. Dr. med., Klinikum St. Georg gGmbH
Other Study IDs: BR-14/06-1; BR-14/06-1
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Incurable Cancer Diseases; Other Incurable Diseases
Keywords: Euthanasia; Assisted Suicide; Assisted Dying; Palliative Care Medicine
MeSH Terms: conditions — Suicide, Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients receiving palliative care due to incurable illness

SUMMARY:
Euthanasia and assisted dying are of growing interest for patients with incurable diseases. The possible methods are widely discussed by patient-societies, physicians, lawyers, theologians and philosophers. During the last years several opinion-polls were conducted with healthy people or medical stuff, but no surveys were conducted to get the attitude of incurable ill patients.

The hypothesis of the investigators' study is: "Palliative Care Medicine is a better option for incurable ill patients than an assisted suicide."

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Incurable illness
* Mental state thet allows to answer a questionnaire

Exclusion Criteria:

* Somnolence
* Low mental state
* Curable disease
* Depression with danger of acute suicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with incurable illness
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-09; Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Patients intention to assisted suicide | up to four weeks after beginning of palliative treatment

CONTACTS AND LOCATIONS:
Overall Officials: Armin R Sablotzki, MD, Principal Investigator — Klinikum St. Georg Leipzig, Clinics of Anesthesiology, Critical Care and Pain Therapy; Matthias Thieme, MD, Study Director — Klinikum St. Georg Leipzig, Clinics of Anesthesiology, Critical Care and Pain Therapy
Locations (1):
- Klinikum St. Georg gGmbH, Leipzig, Saxony, Germany

REFERENCES:
- See also: Homepage of the study site — http://www.sanktgeorg.de